CLINICAL TRIAL: NCT06846073
Title: A Prospective Clinical Study on the Early Combined Use of Dexamethasone Intravitreal Implant and Anti-VEGF in the Treatment of Diabetic Macular Edema (DME) in Naive Patients.
Brief Title: Early Combined Use of Dexamethasone Intravitreal Implant and Anti-VEGF in the Treatment of DME.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ningbo Eye Hospital (Other); Jiaxing Hospital of T.C.M (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0369
Record Dates: First submitted 2024-12-05; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Macular Edema (DME)
Keywords: dexamethasone implant; vascular endothelial growth factor; Corticosteroids; combination therapy; biomarker; best corrected visual acuity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The combination of intravitreal anti-VEGF and dexamethasone implants injections. (Experimental): The patients will receive the combination of intravitreal anti-VEGF and dexamethasone implants injections.
  Interventions: Combination Product: The combination of intravitreal anti-VEGF and dexamethasone implants injections.
- Anti-VEGF injections monotherapy (No Intervention): The patients will receive intravitreal anti-VEGF injections.

INTERVENTIONS:
Combination Product: The combination of intravitreal anti-VEGF and dexamethasone implants injections. — Early combination of intravitreal dexamethasone implant and anti-VEGF injection for the treatment of DME.
  Arms: The combination of intravitreal anti-VEGF and dexamethasone implants injections.

SUMMARY:
The goal of this clinical trial is to learn if the efficacy of dexamethasone implant combined with anti-VEGF superior to anti-VEGF monotherapy in the treatment of DME in Chinese patients. The main questions it aims to answer are:

1. Whether combination therapy improves the best corrected visual acuity at 6 months and 12 months?
2. Does combination therapy improve retinal anatomy better than monotherapy at each time point?

Researchers will compare the combination therapy to the monotherapy to see if dexamethasone implant combined with anti-VEGF will leads to better results.

Participants will:

1. be randomly assigned to one of two groups with equal probability to receive the combination of intravitreal anti-VEGF and dexamethasone implant injections or intravitreal anti-VEGF injections.
2. During the first 3 months, patients in both groups will receive monthly injections of anti-VEGF. In the double protocol group, the first dexamethasone implant injection will be administered simultaneously with the first loading dose of anti-VEGF injections. Between 4 and 12 months, patients will receive intravitreal anti-VEGF injections as needed/pro-re-nata (PRN).
3. Patients will have regular follow-up. Routine examination includes Central retinal thickness (CRT), intraocular pressure (IOP), slit lamp examination, best corrected visual acuity (BCVA) and OCT.

ELIGIBILITY:
Inclusion Criteria:

* Type 1/type 2 diabetes mellitus with good glycaemic control and glycated haemoglobin ≤ 10.0%; DR stage II-III;
* DME with involvement of the central concavity and resulting in the patient's vision loss;
* Central retinal thickness (CRT) ≥250 μm;
* No refractive interval clouding and pupillary constriction affecting fundus examination;
* No Pan-Retinal Photocoagulation treatment within 3 months before enrolment;
* No macular laser treatment in the past or during the follow-up period;
* Good patient cooperation and compliance.

Exclusion Criteria:

* other macular lesions such as macular preexisting membranes, macular schisis, or other causes of macular oedema such as uveitis and central retinal vein occlusion;
* Co-existence of diabetic optic neuropathy;
* Previous intraocular injection therapy such as anti-VEGF drugs or glucocorticoid drugs in the target eye;
* History of vitreoretinal surgery in the target eye;
* A history of uncontrolled stable glaucoma or hypertension, hormonal hypertension in the target eye;
* Aphakic eyes with posterior lens capsule rupture with an anterior chamber IOL (ACIOL), iris or transscleral fixed intraocular IOLs, and patients with posterior lens capsule rupture;
* Pregnant or breastfeeding patients, uncontrolled hypertension within 3 months, cerebrovascular accident or myocardial infarction, uncontrolled diabetes mellitus, or other reasons for not being able to co-operate with the relevant examination;
* Lost visits and data loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Average change in best corrected visual acuity (BCVA) of each group from baseline to the end of month 6. | 6 month.
  BCVA was measured using the log Mar visual acuity chart or the ETDRS visual acuity chart.

SECONDARY OUTCOMES:
Average change in best corrected visual acuity (BCVA) of each group from baseline to month 3, 12. | 3 month and 12 month
  BCVA was measured using the log Mar visual acuity chart or the ETDRS visual acuity chart.
Average change in central retinal thickness (CRT) of each group from baseline to month 3, 6,12. | 3, 6 and 12 month
  Central retinal thickness (CRT) is a measurement of the macula from the internal limiting membrane to the RPE and can be quantified by OCT scans
The proportion of eyes with a 5-letter /10-letter improvement from baseline of BCVA at month 6 and 12. | 6 month and 12 month
  BCVA was measured using the log Mar visual acuity chart or the ETDRS visual acuity chart.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqing Chen, M.D., Study Chair — Eye Center, The Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Eye Center, The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
demographic data, diagnostic results, treatment data, lab test results, follow-up data Etc.